CLINICAL TRIAL: NCT02014805
Title: A Multi-institutional, Randomized Controlled Trial of Postoperative Conformal Radiotherapy for Stage II-III B Type Thymoma
Brief Title: Postoperative Conformal Radiotherapy for Stage II-III B Type Thymoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Hospital (Other Government); 309th Hospital of Chinese People's Liberation Army (Other)
Responsible Party: Principal Investigator, Ye Zhang, Attending physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POCRT
Record Dates: First submitted 2013-12-07; First posted 2013-12-18 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Thymoma
Keywords: postoperative; conformal; radiotherapy; thymoma
MeSH Terms: conditions — Thymoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radiotherapy (Experimental): postoperative conformal radiotherapy for Masaoka stage II-III B type thymoma
  Interventions: Radiation: radiotherapy
- observation (No Intervention): no treatment after radical resection for thymoma

INTERVENTIONS:
Radiation: radiotherapy — postoperative conformal radiotherapy for Masaoka stage II-III B type thymoma
  Arms: radiotherapy

SUMMARY:
The purpose of this study is to determine whether postoperative conformal radiotherapy are effective in the treatment of Masaoka stage II-III B type thymoma.

DETAILED DESCRIPTION:
The role of postoperative radiotherapy in thymoma is controversial. Some retrospective studies were for the radiotherapy, but others were against. However, more inherent biases existed in these trials. Resection, Masaoka stage and pathology were widely accepted as the prognostic factors for thymoma. Furthermore, the frequency of local failure after radical resection was still high in Masaoka stage II-III B type thymoma. With the conformal technique appearing, conformal radiotherapy can escalate the dose without increasing the risk of normal tissue toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75, Zubrod-ECOG-WHO 0-2, the interval of surgery to radiotherapy < 2months, Masaoka stage II-III and WHO B type thymoma

Exclusion Criteria:

* No second primary tumor, no serious comorbidity, no neoadjuvant anticancer treatment, no adjuvant chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2013-07; Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
3 year local control rate | 3 year after the end of all enrollment
  local control: tumor recurrence in the tumor bed 3 year local control rate: number of patients with tumor recurrence in the tumor bed at 3 years

SECONDARY OUTCOMES:
3 year failure-free and overall survival | 3 year after the end of all enrollment
  failure-free survivail: the interval from the surgery and the recurrence within or out the tumor bed overall survival: the interval from the surgery and the death or lost of follow-up

OTHER OUTCOMES:
rate of acute and late radiation toxicity | within 3 year after the end of all enrollment
  toxicity: including the acute radition-induced lung toxicity and the late lung toxicity at 1, 3, 6, 9, 12, 18, 24, 30 and 36 month after radiation or observation
quality of life score | within 3 years after all enrollment
  quality of life: FACT-Lung and EORTC QOL C30 before and after radiation, and at 1, 3, 6, 9, 12, 18, 24, 30, 36 months after radiation or observation

CONTACTS AND LOCATIONS:
Overall Officials: Qinfu Feng, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital, Chineses Academy of Medical Sciences, Beijing, China